CLINICAL TRIAL: NCT00078546
Title: Administration of EBV-Specific Cytotoxic T Lymphocytes Following CD45 Antibody to Patients With EBV Positive Nasopharyngeal Carcinoma
Brief Title: EBV-Specific CTLs Following CD45 Antibody to Patients With Epstein-Barr Virus (EBV) + Nasopharyngeal Carcinoma (NPC)
Acronym: CLANC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Stephen Gottschalk, Associate Professor, Pediatrics Hematology Oncology, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H14214; CLANC; NCT00608257 (obsolete NCT alias)
Record Dates: First submitted 2004-03-01; First posted 2004-03-02 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Nasopharyngeal Cancer; EBV Infections
Keywords: EBV; NASOPHARYNGEAL; CARCINOMA; EBV POSITIVE NASOPHARYNGEAL CARCINOMA
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Epstein-Barr Virus Infections; Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: EBV specific CTL Infusion — One injection at one of the following dose levels
  Dose level I: 2x107/m2 Dose level II: 5x107/m2 Dose level III: 1x108/m2
Biological: Anti CD45 monoclonal antibody — 400ug/kg over 6 to 8 hr for 4 days
  Other Names: YTH 24/54

SUMMARY:
To determine the safety of the combination of CD45 monoclonal antibody (Mab) followed by intravenous injection of EBV specific CTL in patients with nasopharyngeal cancer.

To compare the expansion, persistence and anti-tumor effects of the EBV specific CTL given after CD45 Mab administration with that observed in our first study.

To obtain preliminary information on the safety and response to an extended dosage regimen of EBV-specific CTL in patients, who have stable disease or a partial response after the initial dose of EBV-specific CTL.

DETAILED DESCRIPTION:
Three different doses of CTL will be evaluated: dose level I: 2 x 10e7/m2; dose level II: 5 x 10e7/m2; dose level III: 1 x 10e8/m2

Day 1 YTH 24/54 800ug/kg over 8 hr; Day 2 YTH 24/54 800ug/kg over 8 hr; Day 3 Rest; Day 4-6 CTL Infusion (provided CD45 Mab level <100 ug/ml).

Generation of EBV-specific CTL

After consent on the separate procurement protocol for CTL preparation the patient will donate up to 60-70cc of peripheral blood. 10-20cc of this will be used for the establishment of an EBV transformed lymphoblastoid cell line (EBV-LCL) by infection with virus produced from the B95-8 master cell line. The EBV-LCLs will take approximately four to six weeks to establish. 30-40cc of peripheral blood will be used to generate EBV specific CTLs. The CTL line will be prepared by co-cultivation of the irradiated EBV-LCL with patient PBMC. After establishment, the CTL lines will be checked for identity, phenotype and microbiological culture and cryopreserved prior to administration according to SOPs. The antigen specificity of each CTL line will be determined in cytotoxicity assay and when possible with tetramer reagents.

CD45 monoclonal antibodies

Anti-CD45 is a combination in equal amounts (weight for volume) of two monoclonal antibodies that are directed to non-overlapping epitopes on human CD45. It is a purified, concentrated, and sterile gamma globulin, primarily monomeric IgG, produced from the supernatant of the two rat IgG2b hybridoma clones, YTH 24 and YTH 54. The hybridomas were produced as fusions between splenocytes from DA rats immunized with human leukocytes and the rat myeloma line Y3. The combination of the two MAbs exerts a synergistic effect in vitro on complement-mediated cytotoxicity of white cells and it has been demonstrated to clear almost all passenger leukocytes from donor kidneys before transplant. Anti-CD45 Mabs have been made under cGMP conditions at the Therapeutic Antibody Center at Oxford and at Baylor College of Medicine and will pass the safety tests required by the FDA.

Cell administration

Patients will be pre-medicated with Diphenhydramine 1mg/kg IV (max 50 mg) and Acetaminophen 10mg/kg po (max 650 mg). EBV specific T cells will be given by intravenous injection over 1-10 minutes through either a peripheral or a central line. Outpatients may be treated in the clinic. Monitoring will be undertaken according to institutional standards for administration of blood products with the exception that the injection will be given by a physician. Anti-emetics in appropriate dosage for each patient will be prescribed as necessary. Patients will receive supportive care for acute or chronic toxicity, including blood components or antibiotics, and other intervention as appropriate.

Antibody administration

Patients will be pre-medicated with Diphenhydramine 1mg/kg IV (max 50 mg) and Acetaminophen 10mg/kg po (max 650 mg). 800ug/kg CD45 Mabs will be given as 2 daily intravenous infusions over 8 hours. The antibody aliquot to be infused will arrive in the treatment area hand-carried by the attending physician or appointed designate. The antibody aliquot will be diluted in minimal amounts of normal saline. The resulting solution is stable for 24 hours. The antibody solution is administered by a syringe pump in incremental doses, 0.2-0.8 mg in the first hour and up to 10 mg/hr thereafter, for a total infusion time of a maximum of 6 hrs. A registered nurse and a physician must be readily available.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with EBV positive NPC, in relapse or with primary resistant disease
* Life expectancy of more than 6 weeks.
* No severe intercurrent infection
* Patient, parent/guardian able to give informed consent
* Bilirubin less than 2x normal
* SGOT less than 3x normal,
* Hgb higher than 8.0 g/L
* Creatinine less than 2x normal for age
* Patients should have been off other investigational therapy for one month prior to entry in this study.
* Karnofsky score of over or equal to 50.

Exclusion Criteria:

Due to unknown effects of this therapy on a fetus, pregnant women are excluded from this research. The male partner should use a condom.

Note: Patients who would be excluded from the protocol strictly for laboratory abnormalities can be included at the investigator's discretion after approval by the CCGT Protocol Review Committee and the FDA reviewer.

.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2003-09; Primary Completion 2007-01 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
safety of autologous Epstein Barr Virus (EBV)-specific cytotoxic T-lymphocytes (CTL) in combination with CD45 monoclonal antibody (Mab) in patients with nasopharyngeal cancer | 6 weeks post infustion
obtain information on the expansion, persistence and anti-tumor effects of EBV-specific CTL lines given after lymphodepletion with CD45 Mab in patients with nasopharyngeal cancer | 12 months post infusion
To obtain preliminary information on the safety and response to an extended dosage regimen of EBV-specific CTL in patients, who have stable disease or a partial response after the initial dose of EBV-specific CTL. | 12 months post infusion

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Gottschalk, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Texas Children's Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas

REFERENCES:
- [Derived] Louis CU, Straathof K, Bollard CM, Gerken C, Huls MH, Gresik MV, Wu MF, Weiss HL, Gee AP, Brenner MK, Rooney CM, Heslop HE, Gottschalk S. Enhancing the in vivo expansion of adoptively transferred EBV-specific CTL with lymphodepleting CD45 monoclonal antibodies in NPC patients. Blood. 2009 Mar 12;113(11):2442-50. doi: 10.1182/blood-2008-05-157222. Epub 2008 Oct 29. PMID 18971421